CLINICAL TRIAL: NCT04918043
Title: Raskaudenaikaiset Elintavat ja Etyyliglukuronidin Esiintyminen Mekoniumissa Suomessa
Brief Title: Alcohol Use During Pregnancy in Finland According to Meconium Samples
Acronym: RASMEK21
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hanna Kahila (Other)
Collaborators: Helsinki University Central Hospital (Other); Lastentautien tutkimussäätiö (Unknown)
Responsible Party: Sponsor-Investigator, Hanna Kahila, MD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Other Study IDs: HUS/222/2021
Record Dates: First submitted 2021-05-30; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — meconium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HUCS, NKL: Newborns and their mothers at the Helsinki University Central Hospital maternity ward.

SUMMARY:
Meconium samples are collected anonymously from newborns in Helsinki University Hospital maternity ward. The study tries to to find how many women continue to use alcohol during the second half of the pregnancy. Meconium samples are tested for ethylglucuronide (EtG), a metabolite of ethanol, that accumulates in the meconium. Altogether 1000 samples are taken. The sample results are compared to anonymously answered questionnaire about alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* newborn baby

Exclusion Criteria:

-

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of the newborn babies that are born at the Helsinki University Central hospital maternity ward.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
EtG | Once
  The meconium samples from newborns are tested for ethyl glucuronide using LC-MS/MS mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Kahila, MD, Principal Investigator — HUCS

IPD SHARING:
Plan to Share IPD: Yes
All anonymous IPD will be shared with the modelling source code.
Supporting Information: ICF, Analytic Code
Time Frame: 6 months after the publication
Access Criteria: Scientific study, policy making